CLINICAL TRIAL: NCT05232903
Title: Safety of Stromal Vascular Fraction (SVF) Therapy in Patients With Acute Spontaneous Intracerebral Hemorrhage (SICH): a Phase I Clinical Study
Brief Title: Stromal Vascular Fraction (SVF) Therapy in Patients With Acute Spontaneous Intracerebral Hemorrhage (SICH).
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Dr. Yong Cao, Clinical Professor, Beijing Tiantan Hospital
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SICH-SVF
Record Dates: First submitted 2021-12-06; First posted 2022-02-10 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Spontaneous Intracerebral Hemorrhage
Keywords: Spontaneous intracerebral hemorrhage; Stromal vascular fraction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 SVF dose 0.5 x 10^6/kg Intravenous infusion (IV) (Experimental): Intravenous infusion of stromal vascular fraction (SVF) dose 0.5 x 10^6/kg for 5 participants within 1 month after neurosurgical intracerebral hemorrhage (ICH) evacuation.
  Interventions: Biological: SVF therapy group
- Group 2 SVF dose 1.0 x 10^6/kg Intravenous infusion (IV) (Experimental): Intravenous infusion of stromal vascular fraction (SVF) dose 1.0 x 10^6/kg for next 5 participants within 1 month after neurosurgical intracerebral hemorrhage (ICH) evacuation.
  Interventions: Biological: SVF therapy group
- Group 3 SVF dose 1.5 x 10^6/kg Intravenous infusion (IV) (Experimental): Intravenous infusion of SVF stromal vascular fraction (SVF) dose 1.5 x 10^6/kg for final 5 participants within 1 month after neurosurgical intracerebral hemorrhage (ICH) evacuation.
  Interventions: Biological: SVF therapy group

INTERVENTIONS:
Biological: SVF therapy group — The active treatment is an intravenous injection with the stromal vascular fraction (SVF) harvested from the patient's own fatty tissue.

SUMMARY:
The purpose of this pilot study is to evaluate the safety of stromal vascular fraction (SVF) therapy in patients with spontaneous intracerebral hemorrhage (SICH).

DETAILED DESCRIPTION:
Spontaneous intracerebral hemorrhage (SICH) is a form of brain parenchymal hemorrhage caused by various non-traumatic reasons, resulting in cerebral artery, veins or capillaries rupture. SICH is a common neurological emergency with the characteristics of rapid onset, dangerous conditions, and a high disability and fatality rate. Although the fatality rate has decreased, reflecting the progress of recent medical technologies, most patients still have persistent language or limb movement dysfunction.

Stromal vascular fraction (SVF) is a structural framework in the body's fat tissue, comprising mesenchymal stem cells, white blood cells, red blood cells, endothelial cells, T cells, platelets related cytokines. Previous studies have demonstrated that SVF has favorable therapeutic effects against various diseases regarding different systems, including the motor system, respiratory system, circulatory system, and nervous system, which indicated the treatment potential of SVF in the treatment of SICH.

The overall clinical development strategy of this project is to conduct a Phase I dose-escalation study to evaluate the safety of SVF therapy in patients with SICH. Fifteen patients with SICH will be sequentially assigned to 3 dose groups, and the adverse events (AEs) and serious adverse events (SAEs) will be recorded in a period of 1 year.

ELIGIBILITY:
Inclusion Criteria:

1. Age range: 45~55 years old
2. Acute spontaneous supratentorial ICH documented by head CT with GCS Score between 8-12 inclusive.
3. Stable ICH hematoma volume 60mL or less as measured by ABC2 method based on preoperative CT.
4. Neurosurgical ICH evacuation can be performed within the first 72 h of ICH onset.
5. Ability to provide written personal or surrogate consent.
6. Expectancy life is longer than 12 months.
7. Subject must be available for all specified assessments at the study site through the completion of the study.
8. Determining Organ function according to the following criteria:

1) Aspartate transaminase (AST) ≤2.5×Upper limit of normal 2) Alanine transaminase (ALT) ≤2.5×Upper limit of normal 3) Total bilirubin (T-Bil) ≤1.5×Upper limit of normal 4) Serum albumin (SA) ≥3.0g/dL 5) Absolute neutrophil count（ANC）≥1.5×10^9/L 6) Platelets (PLT) ≥150×10^9/L 7) Hemoglobin (Hb) ≥9.0g/dL 8) Creatine kinase (CK) ≤1.5×Upper limit of normal 9) Serum amylase (AMY) and serum lipase (Lip) are within the normal range

Exclusion Criteria:

1. Secondary ICH related to aneurysm, AVM, trauma, brain tumor, etc.
2. History of epilepsy.
3. History of brain tumor.
4. History of brain trauma.
5. Pre-existing disability defined as a pre-stroke modified Rankin scale >2.
6. Evidence of organ failure.
7. Septicemia with high fever and shock.
8. Positive for any one of hepatitis B surface antigens, e antigens, e antibodies, and core antibodies, hepatitis C virus antibodies, syphilis antibodies, or HIV antibodies positive.
9. Participation in any clinical investigation within 3 months prior to dosing.
10. Suffer from any other clinically significant medical diseases or with evidence of metal disorder.
11. The investigator or sponsor determines that participating in the trial will bring safety risks to the patients.
12. Participated in other stem cell therapy research.
13. History of drug or alcohol abuse in the past year
14. Women who are pregnant, breastfeeding, or planning to become pregnant during the trial
15. Allergic to cattle and pork products.

Ages: 45 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Estimated)
Dates: Start 2022-03-01 (Estimated); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Occurrence of adverse events | 1 year
  Number of adverse events at each Stromal vascular fraction (SVF) dose following infusion.

SECONDARY OUTCOMES:
The changes in stroke-related neurologic deficit | baseline, Month 1, Month 3, Month 6, Month 9, Month 12
  The changes in stroke-related neurologic deficit were measured by the National Institute of Health stroke scale (NIHSS), which ranges from 0 to 45. Higher scores indicate worse neurological function.
The changes in patients' language function | baseline, Month 1, Month 3, Month 6, Month 9, Month 12
  The changes in patients' language function were measured by the Western Aphasia Battery (WAB), which ranges from 0 to 100. Higher scores indicate better language function.
The changes in patients' sensorimotor function | baseline, Month 1, Month 3, Month 6, Month 9, Month 12
  The changes in patients' language function were measured by the Fugl-Meyer Assessment (FMA), which ranges from 0 to 226. Higher scores indicate better language function.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tiantan Hospital Affiliated to Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided